CLINICAL TRIAL: NCT04814407
Title: Developing Novel Circulating Epigenetic Biomarkers for Early Detection of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012096RIPC
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Cell-free DNA; DNA methylation; T cell methylome; cell-free tumor DNA (ctDNA)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung cancer patients: Patients age over 20, with suspected or confirmed diagnosis of lung cancer.
  Interventions: Diagnostic Test: Blood-derived DNA methylation detection
- Indeterminate subjects: Subjects who had indeterminate sub-centimeter pulmonary nodules or ground glass opacities discovered by computed tomography.
  Interventions: Diagnostic Test: Blood-derived DNA methylation detection
- Control subjects: Non-cancer patients including healthy volunteers, chronic inflammatory airway diseases such as chronic obstructive airway disease, asthma, and bronchiectasis, etc.
  Interventions: Diagnostic Test: Blood-derived DNA methylation detection

INTERVENTIONS:
Diagnostic Test: Blood-derived DNA methylation detection — Up to 20 ml of blood will be collected from each subject, and the blood specimen will be processed to isolate plasma cell-free DNA and immune-derived cells (circulating T cells). Circulating methylated tumor/immune signature will then be identified.

SUMMARY:
The investigators aim to identify novel circulating methylated biomarkers for early lung cancer detection as well as to develop new technologies that are clinically applicable with high sensitivity and specificity.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death, accounting for 2.09 million cases in 2018 worldwide. There is a huge demand globally for sensitive and reliable assays to intercept lung cancer at early stages when it can be cured. Past studies have shown that circulating cell-free tumor DNA (ctDNA) shed from tumor cells contains the same mutations and methylation patterns as the original tumor cells. Emerging evidence has indicated the presence of systemic immune dysregulation in cancer patients, and that tumor-reactive T cells carry a distinct molecular profile compared to other bystander cells. Thus, molecular abnormality of ctDNA and tumor-reactive T cells may be one of the early signs that hint the presence of malignancy, and it may serve as a promising target for development of blood-based assays in early lung cancer for its convenience and non-invasiveness as opposed to invasive tumor biopsy, or imaging-based methods that are limited by unsatisfactory sensitivity/specificity.

The investigators aim to identify novel markers for early lung cancer detection as well as to develop new technologies that are clinically applicable with high sensitivity and specificity. The objectives of this proposal are multifaceted: (1) The investigators will generate genome-wide methylation atlas of circulating cell free DNA and of circulating T cells in lung cancer patients vs. non-cancer subjects. (2) The investigators will develop an enriched method to enhance the performance of multiplex droplet digital PCR (ddPCR) technology with increased sensitivity and decreased input DNA requirement. (Enriched methylation-specific droplet digital PCR, EMS-ddPCR) (3) The investigators will develop a single-cell, locus-specific DNA methylation detection system that is bisulfite-free and non-PCR-based. The system can be coupled with flow cytometry or mass cytometry to enable cell-type specific methylation detection. (single-cell, locus-specific methylation detection, scLSM-FACS) (4) The investigators will identify a novel methylation signature consisting of tumor-derived and immune-derived biomarkers for early detection of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suspected or confirmed diagnosis of lung cancer.
* Subjects who had indeterminate sub-centimeter pulmonary nodules or ground glass opacities discovered by computed tomography.
* Non-cancer subjects: including healthy volunteers and chronic inflammatory airway diseases such as chronic obstructive airway disease, asthma, and bronchiectasis, etc.
* Subjects age over 20.

Exclusion Criteria:

* Pregnancy.
* Subjects with HIV infection.
* Unable to or unwilling to give informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Study subjects: Patients with suspected or confirmed diagnosis of lung cancer.
  2. Indeterminate subjects: Subjects who had indeterminate sub-centimeter pulmonary nodules or ground glass opacities discovered by computed tomography.
  3. Control subjects: Non-cancer subjects including healthy volunteers, chronic inflammatory airway diseases such as chronic obstructive airway disease, asthma, and bronchiectasis, etc.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating tumor and immune methylated signature | 1 year
  Genome-wide methylation profile of lung cancer patients and control subjects will be measured both in circulating T cells and cell-free DNA collected from peripheral blood by using Infinium MethylationEPIC BeadChip platform.
Technology development | 1 year
  The investigators will develop enriched methylation-specific droplet digital PCR (EMS-ddPCR) with increased sensitivity and decreased input DNA requirement. The investigators will develop single-cell, locus-specific DNA methylation detection system for flow cytometry (scLSM-FACS) to enable cell-type specific methylation detection.
Technology validation | 1 year
  The investigators will validate the identified circulating methylated signature in patients with indeterminate pulmonary nodules.

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Chen Tsai, M.D., Ph.D, Study Chair — Graduate institute of Toxicology, NTUCM; Department of Internal Medicine, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan